CLINICAL TRIAL: NCT00295373
Title: Phase 4 Clinical Trial to Examine the Role of Rosuvastatin and Exercise Treatment in Modulating Inflammatory Response in Hypercholesterolemic Subjects
Brief Title: Exercise And Rosuvastatin Treatment: Is There an Anti-Inflammatory Synergy?
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Purdue University (Other)
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: 0HQ01; IRB Protocol Ref.#: 0504001888
Record Dates: First submitted 2006-02-21; First posted 2006-02-23 (Estimated); Last update posted 2007-04-20 (Estimated); Status verified 2007-04

CONDITIONS: Nonfamilial Hypercholesterolemia; Physical Inactivity
Keywords: Hypercholesterolemia; Exercise; Statin; Rosuvastatin; TLR4; Inflammation
MeSH Terms: conditions — Sedentary Behavior; Hypercholesterolemia; Motor Activity; Inflammation | interventions — Rosuvastatin Calcium; Exercise

INTERVENTIONS:
Drug: Rosuvastatin
Behavioral: Exercise Training

SUMMARY:
The purpose of this study is to determine whether the effects of rosuvastatin treatment and exercise training can be synergistic, with respect to the innate immune receptor TLR4, markers of systemic inflammation, and stimulated production of inflammatory cytokines, in hypercholesterolemic subjects. It is hypothesized that a rosuvastatin and exercise intervention will synergistically lower measured variables, so as to be anti-inflammatory.

DETAILED DESCRIPTION:
Both statin drugs and exercise training are known to exert anti-inflammatory effects. We found that both high levels of physical activity and an exercise training program reduced markers of inflammation and lowered monocyte Toll-like receptor 4 (TLR4) expression. It has not been determined whether statins exert their anti-inflammatory effects through the toll-like receptors or whether combined statin/exercise treatment will exert synergistic anti-inflammatory effects. Thus, the primary purposes of this study are two-fold: 1) Determine whether rosuvastatin treatment downregulates LPS-induced inflammatory responses, serum hsCRP, and monocyte TLR4 expression in hypercholesterolemic patients; and 2) Determine whether adding exercise training to rosuvastatin treatment induces an anti-inflammatory synergy and further lowers LPS-induced inflammatory response, hsCRP, and TLR4 expression. Thirty two hypercholesterolemic (total cholesterol > 200 mg/dL, LDL > 130 mg/dL) will be randomly divided into two groups: statin (ST) and statin and exercise (ST+E). Sixteen physically active, no-statin subjects will also be recruited as a control group(CON). After baseline blood sampling, ST and ST+E groups will begin a 10-week course of rosuvastatin calcium treatment (10 mg/d) after which a second blood sample will be obtained. The ST+E group will then begin a 10 week (three days per week) combined endurance (20 min at 70% of heart rate reserve) and resistive training (2 sets of 10 upper- and lower-body exercises) program. The ST group will not exercise and both ST+E and ST groups will continue taking their medication, as prescribed. A final blood sample will be taken at the end of this 10-week segment. Blood samples will also be taken from the CON group at 0, 10 and 20 weeks. Monocyte expression of TLR4, CD14 (LPS receptor) and CD16 (monocyte maturation marker) will be assessed using flow cytometry. LPS-stimulated inflammatory cytokine production and serum levels of hsCRP, TNF-a, oxLDL, LDL, HDL, endotoxin, LPS binding protein, and sCD14 will also be measured at each time point (baseline, 10 weeks, 20 weeks). These experiments will allow us to determine whether rosuvastatin downregulates TLR4, an important mediator of inflammation, and whether exercise, known to lower TLR4 expression, can augment the rosuvastatin effects. Regular exercise and statin treatment are known to reduce disease risk, but the benefits of these treatments is infrequently attributed to their anti-inflammatory effects. It is important to document mechanisms of anti-inflammatory action for exercise training and statin treatment and to determining whether these treatments have combined beneficial effects.

ELIGIBILITY:
Inclusion Criteria:

* Nonfamilial hypercholesterolemia
* Total cholesterol >200 mg/dl, LDL >130 mg/dL
* Physical inactivity
* Moderate to low alcohol intake

Exclusion Criteria:

* Liver or kidney disease
* Acute illness or infection
* Use of corticosteroids, ACE inhibitors, platelet aggregating inhibitors, thiazolidinediones, and bis-phosphonates.
* Use of cyclosporine, warfarin, gemfibrozil or other lipid lowering agents
* Regular antacid or aspirin use
* Type I & II diabetes with insulin treatment
* hypothyroidism, and/or renal insufficiency
* Chronic/debilitating osteoarthritis
* Rheumatoid arthritis
* Central or peripheral nervous system disorders
* Anti-depressant medications
* Major affective disorder
* HIV infection or auto-immune disorders
* Use of tobacco products
* unexplained or intended weight loss of > 2 kg during the previous six months
* Surgery within the previous three months

Ages: 40 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48
Dates: Start 2006-02; Study Completion 2007-08 (Estimated)

PRIMARY OUTCOMES:
The following measures will be made at 0, 10 and 20 weeks:
Monocyte cell-surface expression of TLR4, CD14, and CD16
LPS-stimulated whole blood production of IL-6 and TNF-α
Serum levels of hsCRP and TNF-α
Serum levels of Endotoxin LDL, OxLDL, HDL, sCD14, and
Lipopolysaccharide Binding Protein.

SECONDARY OUTCOMES:
Creatine kinase & ALT (0, 5, 10 weeks; rosuvastatin group)
Creatine kinase & ALT (48hrs after 1st and 5th exercise
bout; rosuvastatin + exercise group)

CONTACTS AND LOCATIONS:
Overall Officials: Robert E Hannemann, MD, Principal Investigator — Purdue University; Michael G Flynn, PhD, Study Director — Purdue University
Locations (1):
- Purdue University, West Lafayette, Indiana, United States

REFERENCES:
- [Background] Stewart LK, Flynn MG, Campbell WW, Craig BA, Robinson JP, McFarlin BK, Timmerman KL, Coen PM, Felker J, Talbert E. Influence of exercise training and age on CD14+ cell-surface expression of toll-like receptor 2 and 4. Brain Behav Immun. 2005 Sep;19(5):389-97. doi: 10.1016/j.bbi.2005.04.003. PMID 15963685
- [Background] McFarlin BK, Flynn MG, Campbell WW, Stewart LK, Timmerman KL. TLR4 is lower in resistance-trained older women and related to inflammatory cytokines. Med Sci Sports Exerc. 2004 Nov;36(11):1876-83. doi: 10.1249/01.mss.0000145465.71269.10. PMID 15514501
- [Background] Methe H, Kim JO, Kofler S, Nabauer M, Weis M. Statins decrease Toll-like receptor 4 expression and downstream signaling in human CD14+ monocytes. Arterioscler Thromb Vasc Biol. 2005 Jul;25(7):1439-45. doi: 10.1161/01.ATV.0000168410.44722.86. Epub 2005 Apr 28. PMID 15860745
- See also: Committee on the use of Human Research Subjects at Purdue University — http://www.irb.purdue.edu/